#### INFORMED CONSENT FOR HIV TESTING

Protocol title: Determination of the protective efficacy of the *Pv*CS/Montanide ISA-51 (*Pv*CS.2/M-51) vaccine formulation against controlled infection with *Plasmodium vivax* sporozoites.

| Study location: | Quibdó (Chocó) |
|---|---|
| Principal Investigator: | Sócrates Herrera Valencia, MD |
| Institution: | CENTRO DE ESTUDIOS CLÍNICOS |
| | ASOCLINIC LTDA – IPS |
| <b>Description of the study population:</b> | Adult individuals with and without |
| | previous malaria (naïve and semi-immune |
| | groups) |
| Name of study participant: | |
| Code assigned in the study: | |

**Study code: 2201-3** 

#### 1. Purpose of this consent

You have been invited to undergo **testing for Human Immunodeficiency Virus (HIV) infection** as part of the screening/follow-up examinations for the indicated clinical trial. This test is requested **to protect your safety and** ensure that the study results are interpreted correctly. **Your decision is voluntary and does not affect** your health care or your participation in the main study (except when, according to the protocol criteria, the result is an inclusion/exclusion criterion or requires procedures to be deferred for your safety).

#### 2. What the test involves

- A **venous blood sample** (approx. 5–10 mL) will be taken or, if approved by the protocol, a **rapid** capillary/venous blood **test** will be performed.
- If the screening result is **reactive**, the **confirmatory algorithm** will be performed immediately with supplementary tests validated by the Colombian Ministry of Health.
- The estimated time for delivery of the result and the method of delivery (in person/secure online) will be communicated to you by the study team.

### 3. Expected benefits

- Know your HIV status and, if necessary, access counseling and timely referral to your insurer/IPS for comprehensive care.
- Contribute to **safety** during the clinical trial.

There are no financial benefits for taking this test.

### 4. Risks and discomforts

- Physical: mild pain, bruising, or dizziness associated with venipuncture.
- **Emotional/psychosocial**: anxiety or concern while waiting for or receiving the result.
- **Confidentiality**: minimal risk of unauthorized disclosure, mitigated by strict data protection measures.

You will be offered support and counseling before and after the test.

#### 5. Confidentiality and data protection

- Your data will be treated with **strict confidentiality**, using **codes** instead of your name.
- Access to the information will be restricted to authorized study personnel, regulatory authorities, and the ethics committee when required, preserving your identity.
- The results **will not be shared** with third parties (employers, family members, insurance companies) without your authorization, except where legally required.
- The information will be kept for the time required by the protocol and regulations, in secure repositories.

# **6.** Voluntariness and right to withdraw consent

- You may refuse the test or withdraw your consent at any time, without penalty or loss of benefits to which you are entitled.
- If you decide not to undergo the test and the protocol requires it for safety or scientific reasons, the team will explain the **alternatives** (e.g., deferring procedures, exclusion from the study) and their implications.

# 7. Handling of results

- Negative/Non-reactive: You will be informed of the result, and preventive
  measures will be maintained. You will be reminded of the "immunological
  window" (the period during which a recent infection may not be detected) and, if
  applicable, a repeat test will be scheduled.
- Reactive/Positive: The confirmatory algorithm will be activated. If HIV infection is confirmed:
  - o You will receive individual **post-test counseling**.

- You will be **referred** to your insurer/IPS to begin comprehensive care (including medical evaluation and antiretroviral treatment).
- If the result affects your continued participation in the study due to safety criteria, this will be explained to you, and the appropriate clinical followup will be guaranteed.
- You may indicate with whom you wish to share your result (optional). By default, only you and the study staff who need to use that information for in justified reasons will know it.

#### **8.** Costs and compensation

- The test is free of charge for you.
- No payments are made for taking the test, except for reimbursements/compensation allowed by the protocol (e.g., transportation), when applicable.

## **9.** Alternatives to participation

You can get tested for HIV **outside of the study** at your IPS or through public health programs without affecting your relationship with the research center.

### **10.** Questions, concerns, or complaints

If you have concerns about this consent form, wish to withdraw your authorization, exercise your habeas data rights, or file a complaint, please contact:

- Principal Investigator: Sócrates Herrera Valencia, MD
- Study Coordinator: Myriam Arévalo Ramírez, PhD
- Chair of the Ethics Committee: Ignacio Alberto Concha Eastman, MSc
- Address: Cll 21a Cra 23, Zona Minera, La Virginia, Quibdó, Chocó
- **Telephone numbers:** (57) 317 517 0552 (57) 317 517 0557 310 465 9004.
- Email: sherrera@inmuno.org / marevalo@inmuno.org/
- cei-asoclinic@inmuno.org/alberto.conchaeastman@gmail.com.

# 11. Statements and signatures

**I have read (or had read to me) this HIV testing consent form.** I have had the opportunity to ask questions and all of them have been answered clearly. I understand the purpose, risks, benefits, confidentiality, and my rights. **I** voluntarily **authorize** the HIV test to be performed as described.

I authorize my results to be shared with (optional):

| [ ] No one (only me) |
|---|
| [ ] My treating physician for the study |
| [ ] My IPS/insurer |
| [ ] Other: |
| I authorize the study team to contact me to deliver the results by: |
| [ ] In person |
| [ ] Phone call |
| [ ] Secure email/patient portal |
| Do I authorize the retention of a sample aliquot exclusively for the repetition/confirmation of this test, in accordance with current regulations? |
| [ ] Yes [ ] No |
| Participant's name: |
| Identification document: |
| Participant's signature: |
| Date: |
| Witness signature (if applicable): |
| Witness signature: |
| Date: |
| Signature of the investigator or authorized delegate: |
| Date: |